CLINICAL TRIAL: NCT05324761
Title: Pregabalin Versus Gabapentin Efficacy in the Management of Neuropathic Pain Associated With Failed Back Surgery Syndrome
Brief Title: Management of Pain Associated With Failed Back Surgery Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Kindy College of Medicine (Other)
Responsible Party: Principal Investigator, Laith Thamer Al-Ameri, assistant Professor, Al-Kindy College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13 Al-KindyCM
Record Dates: First submitted 2022-03-20; First posted 2022-04-12 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Failed Back Surgery Syndrome
Keywords: Pregabalin; Gabapentin; neuropathic pain; spine surgery
MeSH Terms: conditions — Failed Back Surgery Syndrome; Neuralgia | interventions — Pregabalin; Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin (Active Comparator): A dose of 75 mg of Pregabalin twice daily for one month will be prescribed to each patient enrolled this study arm
  Interventions: Drug: Pregabalin 75mg
- Gabapentin (Active Comparator): A dose of 300 mg of Gabapentin twice daily for one month will be prescribed to each patient enrolled this study arm
  Interventions: Drug: Gabapentin 300mg

INTERVENTIONS:
Drug: Pregabalin 75mg — Each patient complaining of pain associated with spine surgery who is randomly enrolled this arm of the study and start the specific medication of the arm with the recommended dose and duration for a period of one month, patient will be followed regularly regarding compliance to doses and to register any side effect.
  Arms: Pregabalin
Drug: Gabapentin 300mg — Each patient complaining of pain associated with spine surgery who is randomly enrolled this arm of the study and start the specific medication of the arm with the recommended dose and duration for a period of one month, patient will be followed regularly regarding compliance to doses and to register any side effect.
  Arms: Gabapentin

SUMMARY:
Neuropathic pain is a common complication following different types of spine surgery making negative impact on health, along with life style changes and management, many neurologist prescribed either Pregabalin or Gabapentin to manage this condition with overall good results.

our study aims to evaluate the efficacy of Pregabalin and Gabapentin in the management of this condition and to compare between them

ELIGIBILITY:
Inclusion Criteria:

* Patients with Previous spine surgery and subsequent chronic back pain

Exclusion Criteria:

* Patients with connective tissue diseases
* Patients with psychiatric illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Efficacy in Neuropathic pain management | outcome will be assessed one month after the initiation of medication
  Visual analogue scale pain, minimum score is 0, maximum is 10, the higher ther score the more severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Laith Al-Ameri, Study Director — University of Baghdad - Al-Kindy College of Medicine
Locations (1):
- Laith Thamer Al-Ameri, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No